CLINICAL TRIAL: NCT05089682
Title: Morpheus - Manipulating and Optimizing Brain Rhythms for Enhancement of Sleep
Brief Title: Manipulating and Optimizing Brain Rhythms for Enhancement of Sleep
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Unable to enroll subjects due to COVID and complexity of study.
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Gregory Worrell, Principal Investigator, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 19-001216
Record Dates: First submitted 2021-08-16; First posted 2021-10-22 (Actual); Results first posted 2023-11-01 (Actual); Last update posted 2023-11-01 (Actual); Status verified 2023-10

CONDITIONS: Neurological Disease; Parkinson Disease; Epilepsy
Keywords: Deep Brain Stimulation
MeSH Terms: conditions — Nervous System Diseases; Parkinson Disease; Epilepsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Deep Brain Stimulation (DBS) system (Experimental): Subjects with existing DBS systems implanted for neurological disease (e.g., Parkinson's, pain, epilepsy) will have targeted stimulation patterns during specific stages of sleep using their existing DBS device.
  Interventions: Device: DBS Stimulation during sleep

INTERVENTIONS:
Device: DBS Stimulation during sleep — Open and closed-loop electrical modulation triggered and based on ongoing sleep staging by researcher as well as automated closed-loop algorithm for stimulation.

SUMMARY:
The aim of this study is to investigate whether researchers can improve sleep quality in patients with deep brain stimulators by delivering targeted stimulation patterns during specific stages of sleep.

ELIGIBILITY:
Inclusion Criteria:

* DBS in one of the defined nuclei of interest during the period of the study
* Be willing and able to give written and oral informed consent
* Ability to complete all required study procedures including travelling to Mayo Clinic and staying overnight
* All women of childbearing potential and women who have been amenorrheic for less than 1 year must practice effective contraception during the study. This includes a barrier method such as condom or diaphragm with spermicide; barrier intrauterine device (IUD) or abstinence.

Exclusion Criteria:

* Cognitive impairment (judged by the clinician taking consent as not having sufficient mental capacity to understand the study and its requirements). This is including anyone who, in the opinion of the clinician taking consent is unlikely to retain sufficient mental capacity for the duration of their involvement in the study.
* Patients with any other medical condition that would interfere with study conduct or make it unsafe for them to participate
* Pregnancy test positive.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2021-06-22 (Actual); Primary Completion 2021-12-18 (Actual); Study Completion 2021-12-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gregory Worrell, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Deep Brain Stimulation (DBS) System
Started | 4
Completed | 2
Not Completed | 2
Not completed — Withdrawal by Subject | 2

BASELINE CHARACTERISTICS:
Arm/Group | Deep Brain Stimulation (DBS) System
Number analyzed (Participants) | 4
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.75 (5.25)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 4
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 4
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 4

OUTCOME MEASURES:

1. Primary Outcome: Participants to Complete Study
Description: Total number of participants to complete all scheduled study activities
Time Frame: Through study completion, approximately 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Deep Brain Stimulation (DBS) System
Number analyzed (Participants) | 4
Participants | 2

2. Secondary Outcome: Total Sleep Time
Description: Length of sleep time reported in minutes
Time Frame: Baseline, post-intervention (approximately 1 night)
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Deep Brain Stimulation (DBS) System
Number analyzed (Participants) | 2
minutes
  Baseline | 497 (38.18)
  High Frequency Stimulation (40 Hz - 250 Hz) | 490 (26.87)
  Low Frequency Stimulation (2 Hz - 40 Hz) | 432.5 (43.14)

3. Secondary Outcome: Psychomotor Vigilance Test
Description: Measures reaction time (milliseconds) by asking subjects to press a button on an electronic device as soon as a light appears (every few seconds for 10 minutes).
Time Frame: Baseline, post-intervention (approximately 1 night)
Measure: Mean (Standard Deviation); unit: milliseconds
Arm/Group | Deep Brain Stimulation (DBS) System
Number analyzed (Participants) | 2
milliseconds
  Baseline | 388.20 (50.12)
  High Frequency Stimulation (40 Hz - 250 Hz) | 422.83 (72.61)
  Low Frequency Stimulation (2 Hz - 40 Hz) | 392.72 (44.22)

4. Secondary Outcome: Karolinska Sleepiness Scale
Description: Measures subjective level of tiredness at a particular time during the day using a 9-point scoring scale of 1 = extremely alert, 3 = alert, 5 = neither alert nor sleepy, 7 = sleepy - but no difficulty remaining awake, and 9 = extremely sleepy - fighting sleep.
Time Frame: Baseline, post-intervention (approximately 1 night)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Deep Brain Stimulation (DBS) System
Number analyzed (Participants) | 2
score on a scale
  Baseline | 3.83 (1.60)
  High Frequency Stimulation (40 Hz - 250 Hz) | 3.67 (1.21)
  Low Frequency Stimulation (2 Hz - 40 Hz) | 4.17 (1.60)

5. Secondary Outcome: Latency to Sleep Onset
Description: Time in minutes from beginning of study to the first stage of sleep
Time Frame: Baseline, post-intervention (approximately 1 night)
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Deep Brain Stimulation (DBS) System
Number analyzed (Participants) | 2
minutes
  Baseline | 19 (14.14)
  High Frequency Stimulation (40 Hz - 250 Hz) | 14 (0)
  Low Frequency Stimulation (2 Hz - 40 Hz) | 9.5 (10.61)

6. Secondary Outcome: Latency to Rapid Eye Movement (REM) Sleep
Description: Time in minutes from beginning of sleep to first REM sleep onset.
Time Frame: Baseline, post-intervention (approximately 1 night)
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Deep Brain Stimulation (DBS) System
Number analyzed (Participants) | 2
minutes
  Baseline | 149 (86.27)
  High Frequency Stimulation (40 Hz - 250 Hz) | 114.5 (58.69)
  Low Frequency Stimulation (2 Hz - 40 Hz) | 76.5 (47.38)

7. Secondary Outcome: Number of Sleep Cycles
Description: Total number of sleep cycles defined as switches of non-rapid eye movement (NREM) and rapid eye movement (REM) sleep.
Time Frame: Baseline, post-intervention (approximately 1 night)
Measure: Mean (Standard Deviation); unit: number of sleep cycles
Arm/Group | Deep Brain Stimulation (DBS) System
Number analyzed (Participants) | 2
number of sleep cycles
  Baseline | 4 (2.83)
  High Frequency Stimulation (40 Hz - 250 Hz) | 4 (1.41)
  Low Frequency Stimulation (2 Hz - 40 Hz) | 4 (1.41)

8. Secondary Outcome: Number of Awakenings Per Night
Description: Total number of awakenings during night
Time Frame: Baseline, post-intervention (approximately 1 night)
Measure: Mean (Standard Deviation); unit: number of awakenings
Arm/Group | Deep Brain Stimulation (DBS) System
Number analyzed (Participants) | 2
number of awakenings
  Baseline | 28.5 (2.12)
  High Frequency Stimulation (40 Hz - 250 Hz) | 27 (1.41)
  Low Frequency Stimulation (2 Hz - 40 Hz) | 20 (1.41)

ADVERSE EVENTS:
Time Frame: Adverse events were collected from baseline to end of study participation for a total of approximately 4 days on all participants.
Arm/Group | Deep Brain Stimulation (DBS) System
All-Cause Mortality (participants affected / at risk) | 0/4
Serious Adverse Events (participants affected / at risk) | 0/4
Other Adverse Events (participants affected / at risk) | 0/4

LIMITATIONS AND CAVEATS:
This study was terminated due to inability to enroll subjects due to COVID and complexity of study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-01-27): https://cdn.clinicaltrials.gov/large-docs/82/NCT05089682/Prot_SAP_000.pdf
  • Informed Consent Form (2023-01-13): https://cdn.clinicaltrials.gov/large-docs/82/NCT05089682/ICF_001.pdf